CLINICAL TRIAL: NCT03943979
Title: Pilot Study of an Intervention Involving Cognitive Training and Transcranial Direct-current Stimulation (tDCS) in Morbidly Obese Subjects
Brief Title: Pilot Study of an Intervention Involving Cognitive Training and tDCS in Morbidly Obese Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Collaborators: Neuroelectrics Corporation (Industry)
Responsible Party: Principal Investigator, Albert Goday Arno, Medical doctor, Parc de Salut Mar
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IMIMFTLC/EC-TDCS OM
Record Dates: First submitted 2018-06-14; First posted 2019-05-09 (Actual); Last update posted 2019-05-09 (Actual); Status verified 2019-05

CONDITIONS: Obesity, Morbid; Obesity (BMI > 35) and Diabetes Mellitus; Obesity (BMI > 35) and High Blood Pressure; Obesity (BMI > 35) and Dyslipemia
MeSH Terms: conditions — Obesity, Morbid; Obesity; Diabetes Mellitus; Hypertension | interventions — Cognitive Training; Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Active Control group: Subjects will receive CT and sham tDCS during four consecutive days.
  Active group: Subjects will receive CT and active tDCS during four consecutive days.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The difference between the two groups is the tDCS therapy. To mask this difference, the duration time of the session will be the same under both conditions but a standard Sham tDCS protocol will be used for the Active Control group. That is, a 3-sec ramp-up and ramp-down current stimulation, so the subject perceives the current just like the real tDCS, but it is not strong nor durable enough to have any effect on the neuronal activity.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Control group (Sham Comparator): This group will receive CT and sham tDCS each day, for four days.
  Interventions: Other: Cognitive Training
- Active group (Active Comparator): This group will receive both CT and tDCS, each day, for four days.
  Interventions: Other: Cognitive Training; Device: transcranial Direct-Current Stimulation (tDCS)

INTERVENTIONS:
Other: Cognitive Training — Cognitive Training (CT): 4 consecutive days, 30-45 min session involving 5 different tasks designed to train executive functions and attention, available at the Guttmann Neuropersonaltrainer platform (computerized cognitive training tool certified by the Spanish Agency for Medicines and Health Products as a Class I Health Product). The difficulty level of all the tasks was automatically adjusted on a trial-by-trial basis for both Active and Active Control conditions.
Device: transcranial Direct-Current Stimulation (tDCS) — tDCS: 4 consecutive days, 20 min session, delivered through multichannel tDCS (Starstim, Neuroelectrics), with an excitatory target over the r-dlPFC, and an inhibitory target on the contralateral lobe (l-dlPFC). The positioning of the multichannel tCS (electrode location and currents) was solved using the Stimweaver (Ruffini 2013). The resulting tCS montage employed 8 gelled Ag/AgCl electrodes of π cm2 size (Pistim, Neuroelectrics) placed at AF3(-1093uA), AF4 (1178uA), F3 (-1161uA), F4 (1104uA), F7 (-414uA), F8 (530uA), FC5 (1189uA), FC6 (-1332uA).
  Arms: Active group

SUMMARY:
The study aims to: 1) investigate the effects of cognitive training (CT) and combined CT and transcranial direct current stimulation (tDCS) on food intake and 2) to further understand its neuropsychological and neurophysiological basis (i.e. EEG) as well as its impact in endocannabinoids (EC) in a sample of morbidly obese patients seeking for a gastric bypass surgery

DETAILED DESCRIPTION:
The study will explore the impact of a 4-day intervention with either CT (Active control condition) or CT+tDCS (Active condition) stimulation on food intake in a sample of morbidly obese patients, as measured by dietary assessments the week before, during and the week after the intervention. Additionally, to further understand the neuropsychological and neurophysiological basis of its impact, measures of executive function and attention performance and EEG recordings, respectively, will be collected. Furthermore, we will explore the effect of the intervention on endocannabinoids previously related to eating behaviour.

The Active Control condition will receive sham stimulation together with CT, through a computerized cognitive training platform (Guttmann NeuropersonalTrainer), including different tasks with designed to train executive functions and attention. Each session will last approximately 30-40 min.

The Active condition will receive tDCS stimulation (20 min, multichannel with an excitatory target over the r-dlPFC) together with CT (same as for the Active Control condition).

Participants will undergo a basal (the week before intervention) and a post treatment assessments (the day after finishing the intervention) that will include medical history, blood testing, anthropometric measures, a cognitive assessment battery and a 4-day dietary assessment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of both gender, aged between 18 and 60 years-old
* Having a BMI > 40 kg/m2 or having a BMI>35 and suffering from diabetes mellitus, HBP or LDP.
* Obesity conventional treatment failure
* Wish of bariatric surgery
* Accepting the study and signing the Informed Consent

Exclusion Criteria:

* Do not meet inclusion criteria
* Being left-handed
* Using a pacemaker or deep cerebral stimulation device
* Having a psychiatric disease or serious disease
* Neurologic condition or learning issue or mental backwardness that could affect cognitive function
* Use of psycho-stimulating medicines and/or drugs, abuse or dependance to a psychoactive substance (or during the last 6 months)
* Dependance to alcohol or/and drugs (excepted from nicotina)
* In treatment with benzodiazepines, antipsychotics, tricyclic antidepressants or topiramate, started in the last month
* History of psychiatric disorders treated with lithio carbonate.
* Cutaneous lesion on the area of using of electrodes
* Contact allergy to material used in the used devices.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2016-02-25 (Actual); Primary Completion 2017-05-26 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
Change in food intake | 4 consecutive days during the week before starting the treatment; 4 consecutive days during the week of treatment;
  Changes in food consumption (medium kcal intake ) from baseline to the end of the treatment measured by 4-day food registers during the week before starting the treatment and during the 4 days of treatment. The dietary records were checked by a nutritionist and analyzed through the software PCN Pro 1.0.
Stability of changes in food intake | 4 consecutive days during the week before starting the treatment and 4 consecutive days during the week after finishing the treatment
  Changes in food consumption (medium kcal intake ) from baseline to the follow-up assessment measured by 4-day food registers during the week before starting the treatment and the week after finishing the treatment. The dietary records were checked by a nutritionist and analyzed through the software PCN Pro 1.0.

SECONDARY OUTCOMES:
Change in electroencephalogram (EEG) power and coherence | Every training session (4 consecutive days), 3 minutes before starting the training session and 3 minutes after finishing the training.
  EEG was recorded before and after tCS/sham using a Starstim device (Neuroelectrics), same electrode positions as for the stimulation with a sampling frequency of 500 S/s . Electrode impedance: below 10kΩ; electrical reference placed at the right earlobe. EEG data was analyzed offline by means of customized Matlab code (MathWorks Inc. Natick, MA, USA). Data was split into 1s non-overlapping epochs (epochs with amplitudes >50 μV were rejected). EEG-metrics extracted: EEG-power and coherence. To compute EEG power, the power spectral density (PSD) was estimated for each epoch. Band Power was computed for the bands θ=[4,8 Hz], α=[8,13 Hz] β=[13,25 Hz], γ=[30, 45 Hz] and broadband=[4-45Hz] by integrating the PSD within the band frequency limits. Functional connectivity was estimated by means of coherence by the Welch method averaged over all electrodes. Frontal asymmetry (FA) computed as follows: log(avg(AF4 F4 F8 FC6))-log(avg(AF3 F3 F7 FC5); FA<0 reflects dominance of left-hemisphere
Change in Body Mass Index (BMI) | One day during the week before starting the training (pre-treatment) and the 1 day after finishing the treatment (post-treatment)
  Change in BMI. BMI calculation: body weight divided by the square of the body height (expressed in units of kg/m2). Weight and height measures were taken by a nurse.
Change in endocannabinoids (and related compounds) plasmatic concentrations. | One day during the week before starting the training (pre-treatment) and the 1 day after finishing the treatment (post-treatment)
  Change in endocannabinoids and related compounds (acylglycerols and fatty acid N-acylethanolamides) as measured in plasmatic concentrations and quantified by LC/MS-MS by a previously validated method (Pastor et al. 2014).
Change in hormonal measurements : Leptin and adiponectin plasmatic/serum concentrations | One day during the week before starting the training (pre-treatment) and the 1 day after finishing the treatment (post-treatment)
  Measurement of change in hormones regulating the appetite and energic homeostasis of secretion in fatty tissues.
Change in neuropsychological test: Intra-extra dimension (IED-CANTAB Cambridge Cognition) | One day during the week before starting the training (pre-treatment) and the 1 day after finishing the treatment (post-treatment)
  Executive functions: flexibility
Change in neuropsychological test: Stroop Colours and Words test (SCWT, Golden C.J., 1978; Stroop, 1935) | One day during the week before starting the training (pre-treatment) and the 1 day after finishing the treatment (post-treatment)
  Executive functions: inhibition
Change in neuropsychological test: Iowa Gambling Task (IGT, Bechara et al., 1994, 2002) | One day during the week before starting the training (pre-treatment) and the 1 day after finishing the treatment (post-treatment)
  Executive functions: decision-making, risky behaviour.
Change in neuropsychological test: Spatial Span (SSP; CANTAB Cambridge Cognition) | One day during the week before starting the training (pre-treatment) and the 1 day after finishing the treatment (post-treatment)
  Executive functions: working memory
Change in neuropsychological test: Stockings of Cambridge (SOC; CANTAB Cambridge Cognition) | One day during the week before starting the training (pre-treatment) and the 1 day after finishing the treatment (post-treatment)
  Executive functions: planning
Change in neuropsychological test: Conners Continuous Performance Test (CPT, Conners & MHS Staff, 2000) | One day during the week before starting the training (pre-treatment) and the 1 day after finishing the treatment (post-treatment)
  Executive functions: Attention
Change in neuropsychological test: Simple Reaction Time (SRT; CANTAB Cambridge Cognition) | One day during the week before starting the training (pre-treatment) and the 1 day after finishing the treatment (post-treatment)
  Executive functions: Attention
Change in neuropsychological test:Symbol digit modalities test (SDMT; Smith A. 1982). | One day during the week before starting the training (pre-treatment) and the 1 day after finishing the treatment (post-treatment)
  Executive functions: Attention and Processing speed

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Alonso-Alonso M. Translating tDCS into the field of obesity: mechanism-driven approaches. Front Hum Neurosci. 2013 Aug 27;7:512. doi: 10.3389/fnhum.2013.00512. eCollection 2013. PMID 23986687
- [Background] Barr MS, Fitzgerald PB, Farzan F, George TP, Daskalakis ZJ. Transcranial magnetic stimulation to understand the pathophysiology and treatment of substance use disorders. Curr Drug Abuse Rev. 2008 Nov;1(3):328-39. doi: 10.2174/1874473710801030328. PMID 19630729
- [Background] Boivin JR, Piscopo DM, Wilbrecht L. Brief cognitive training interventions in young adulthood promote long-term resilience to drug-seeking behavior. Neuropharmacology. 2015 Oct;97:404-13. doi: 10.1016/j.neuropharm.2015.05.036. Epub 2015 Jun 9. PMID 26066577
- [Background] Conti CL, Moscon JA, Fregni F, Nitsche MA, Nakamura-Palacios EM. Cognitive related electrophysiological changes induced by non-invasive cortical electrical stimulation in crack-cocaine addiction. Int J Neuropsychopharmacol. 2014 Sep;17(9):1465-75. doi: 10.1017/S1461145714000522. Epub 2014 Apr 28. PMID 24776374
- [Background] Corbett A, Owen A, Hampshire A, Grahn J, Stenton R, Dajani S, Burns A, Howard R, Williams N, Williams G, Ballard C. The Effect of an Online Cognitive Training Package in Healthy Older Adults: An Online Randomized Controlled Trial. J Am Med Dir Assoc. 2015 Nov 1;16(11):990-7. doi: 10.1016/j.jamda.2015.06.014. PMID 26543007
- [Background] Ditye T, Jacobson L, Walsh V, Lavidor M. Modulating behavioral inhibition by tDCS combined with cognitive training. Exp Brain Res. 2012 Jun;219(3):363-8. doi: 10.1007/s00221-012-3098-4. Epub 2012 Apr 25. PMID 22532165
- [Background] Gluck ME, Alonso-Alonso M, Piaggi P, Weise CM, Jumpertz-von Schwartzenberg R, Reinhardt M, Wassermann EM, Venti CA, Votruba SB, Krakoff J. Neuromodulation targeted to the prefrontal cortex induces changes in energy intake and weight loss in obesity. Obesity (Silver Spring). 2015 Nov;23(11):2149-56. doi: 10.1002/oby.21313. PMID 26530931
- [Background] Goldman RL, Borckardt JJ, Frohman HA, O'Neil PM, Madan A, Campbell LK, Budak A, George MS. Prefrontal cortex transcranial direct current stimulation (tDCS) temporarily reduces food cravings and increases the self-reported ability to resist food in adults with frequent food craving. Appetite. 2011 Jun;56(3):741-6. doi: 10.1016/j.appet.2011.02.013. Epub 2011 Feb 23. PMID 21352881
- [Background] Grall-Bronnec M, Sauvaget A. The use of repetitive transcranial magnetic stimulation for modulating craving and addictive behaviours: a critical literature review of efficacy, technical and methodological considerations. Neurosci Biobehav Rev. 2014 Nov;47:592-613. doi: 10.1016/j.neubiorev.2014.10.013. PMID 25454360
- [Background] Jauch-Chara K, Kistenmacher A, Herzog N, Schwarz M, Schweiger U, Oltmanns KM. Repetitive electric brain stimulation reduces food intake in humans. Am J Clin Nutr. 2014 Oct;100(4):1003-9. doi: 10.3945/ajcn.113.075481. Epub 2014 Aug 6. PMID 25099550
- [Background] Juarascio AS, Manasse SM, Espel HM, Kerrigan SG, Forman EM. Could training executive function improve treatment outcomes for eating disorders? Appetite. 2015 Jul;90:187-93. doi: 10.1016/j.appet.2015.03.013. Epub 2015 Mar 14. PMID 25777264
- [Background] Sauvaget A, Trojak B, Bulteau S, Jimenez-Murcia S, Fernandez-Aranda F, Wolz I, Menchon JM, Achab S, Vanelle JM, Grall-Bronnec M. Transcranial direct current stimulation (tDCS) in behavioral and food addiction: a systematic review of efficacy, technical, and methodological issues. Front Neurosci. 2015 Oct 9;9:349. doi: 10.3389/fnins.2015.00349. eCollection 2015. PMID 26500478